CLINICAL TRIAL: NCT05591066
Title: The Patient and Family Centered I-PASS LISTEN Study: Language, Inclusion, Safety, and Teamwork for Equity Now
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Pediatric Research in Inpatient Settings (Unknown)
Responsible Party: Principal Investigator, Alisa Khan, Pediatric Hospitalist/Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB-P00042876
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Communication
Keywords: Family Centered Rounds; Patient Safety; Errors; Limited English Proficiency; Health Disparities; Adverse Events; Patient Experience; Family Engagement; Interprofessional Communication; Language Barriers
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Unstructured communication during rounds and unstandardized interpretation at provider discretion.
- PFC I-PASS Intervention (Experimental): Patient and Family-Centered I-PASS is a bundle of communication interventions to improve the quality of information exchange between physicians, nurses, and families, and to better integrate families into all aspects of daily decision making in hospitals. The intervention included a health literacy-informed, structured communication framework for family-centered rounds; written rounds summaries for families; a training and learning program; and strategies to support teamwork and implementation.
  Interventions: Behavioral: PFC I-PASS Intervention
- PFC I-PASS+ Intervention (Experimental): PFC I-PASS+ includes all parts of PFC I-PASS plus having interpreters on and after rounds and training doctors about communication and cultural humility.
  Interventions: Behavioral: PFC I-PASS+ Intervention

INTERVENTIONS:
Behavioral: PFC I-PASS Intervention — Patient and Family-Centered I-PASS is a bundle of communication interventions to improve the quality of information exchange between physicians, nurses, and families, and to better integrate families into all aspects of daily decision making in hospitals. The intervention included a health literacy-informed, structured communication framework for family-centered rounds; written rounds summaries for families; a training and learning program; and strategies to support teamwork and implementation.
  Arms: PFC I-PASS Intervention
Behavioral: PFC I-PASS+ Intervention — PFC I-PASS+ builds on PFC I-PASS to make it better and focus on the special needs of patients who speak languages other than English. PFC I-PASS+ includes all parts of PFC I-PASS plus having interpreters during and after rounds, cultural humility training, and provider communication skills training.
  Arms: PFC I-PASS+ Intervention

SUMMARY:
In 2014, a team of parents, nurses, and physicians created Patient and Family Centered I-PASS (PFC I-PASS), a bundle of communication interventions to improve the quality of information exchange between physicians, nurses, and families, and to better integrate families into all aspects of daily decision making in hospitals. PFC I-PASS changed how doctors and nurses talk to patients and families on rounds when they're admitted to the hospital. (Rounds are when a team of doctors visit patients every morning to do a checkup and make a plan for the day.) Rounds used to happen in a way that left out patients and families. Doctors talked at, not with patients, used big words and medical talk, and left nurses out. PFC I-PASS changed rounds by including families and nurses, using simple non-medical words, and talking in an organized way so nothing is left out. When PFC I-PASS was put in place in 7 hospitals, patients had fewer adverse events and better hospital experience. But it didn't focus on how to talk with patients with language barriers. This project builds upon upon PFC I-PASS to make it better and focus on the special needs of patients who speak languages other than English. This new intervention is known as PFC I-PASS+. PFC I-PASS+ includes all parts of PFC I-PASS plus having interpreters on and after rounds and training doctors about communication and cultural humility. The study team will now conduct a stepped-wedge cluster randomized trial to compare the effectiveness of PFC I-PASS+ and PFC I-PASS to usual care at 8 hospitals.

DETAILED DESCRIPTION:
Hospitalized patients who use languages other than English (LOE, Box 1) for care are at high risk for adverse events (AEs) due to communication failures. These failures include underutilizing safety-promoting strategies, such as certified interpreters, high-reliability structured communication, and family engagement. Patients using LOE also face individual bias from providers (eg, assuming lower intelligence based on accent) and systemic bias from systems not designed to meet their needs (eg, hospitals failing to invest in translation services), which lead to safety risks and poorer health. Patients using LOE also face intersectional bias based on race and ethnicity and other characteristics.

With PCORI's support, the investigators developed a structured communication intervention-Patient and Family Centered I-PASS (PFC I-PASS)-to improve family engagement on rounds that led to a 38% reduction in preventable AEs and improved hospital experience. In the subset of patients/families with language barriers, AEs and hospital experience improved further. However, sites struggled with how to implement PFC I-PASS in patients using LOE for care. Disparities in family engagement in patients using LOE for care persisted and interpreter use varied. The investigators have bolstered PFC I-PASS with evidence-based strategies, including standardized use of certified in-person and video interpreters during and after rounds, cultural humility training, and provider communication skills training (PFC I-PASS+).

The overall goal of this project is to compare the effectiveness of PFC I-PASS+ and PFC I-PASS vs usual care (unstructured communication and unstandardized interpretation at provider discretion) in a population of hospitalized children using LOE (PCORI populations of interest). To pursue this goal, the investigators will conduct a multicenter Hybrid Type I effectiveness trial. The investigators will randomize 4 sites to PFC I-PASS+ and 4 site to PFC I-PASS, using a Stepped Wedge Cluster Randomized Trial (SW-CRT) design to compare the effectiveness of PFC I-PASS and I-PASS+ vs usual care. The investigators will compare safety, experience, discrimination, and communication using gold standard systematic safety surveillance and patient/ family-reported measures. Our primary aim is to test the hypothesis that among patients using LOE for care, both PFC I-PASS+ and PFC I-PASS, vs usual care, will improve: AE rates, patient/family experience of provider communication and experience of discrimination, and communication openness, and frequency of patient-provider communications using interpreters.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the pediatric inpatient study units of participating hospitals
* Patients themselves who are age 13 and up (if they provide assent and their parent or guardian gives permission)*
* Parents/caregivers of patients of all ages who speak English, Arabic, Armenian, Bengali, Chinese (Mandarin and Cantonese), Karen, Korean, Nepali, Quiche, Spanish, Somali, and Vietnamese (and/or other languages if resources allow)
* Nurses working on these units
* Residents working on these units
* Medical and nursing students working on these units
* Hospital leaders working at these hospitals
* *Note for Consenting: Patients (13-18yo) who are in state custody and assent for themselves to complete surveys but lack legal guardian/caregiver present to offer consent are not being approached to complete surveys. These patients may still be enrolled in the study but not consented to complete patient-facing forms.

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14400 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event Rates | 24 months (including usual care and intervention implementation data collection which will happen sequentially) per site (8 sites total)
  Chart review, self-reported by staff and patients/families, and hospital incident reports

SECONDARY OUTCOMES:
Patient/Family Experience with Care Questionnaire | 24 months (including usual care and intervention implementation data collection which will happen sequentially) per site (8 sites total)
  Self-reported by patients/families prior to discharge, based on a previously developed experience survey and modified Child HCAHPS items. Most items are scored on a 5-point Likert scale with higher numbers being better. Top-box (5 or 5 out of 5 scores) will be analyzed.
Patient/Family Experience of Discrimination (Discrimination In Medical Settings Scale) | 24 months (including usual care and intervention implementation data collection which will happen sequentially) per site (8 sites total)
  Self-reported by patients/families prior to discharge through the Discrimination in Medical Settings (DMS) Scale, which is a modified version of the Everyday Discrimination Scale (EDS) adapted to medical settings. The EDS is one of the most utilized self-reported measures of discrimination and is validated across multiple populations. The 7-item DMS Scale has excellent convergent validity and discriminant validity, internal consistency, test-retest reliability, and is used in a variety of clinical conditions. Items include whether patients are treated with less courtesy, less respect, receive poorer services; whether doctor or nurse acts as if patient is not smart, better than patient, or does not listen to patient. Responses were assessed with a 5-point Likert scale (1-never, 2-rarely, 3-sometimes, 4-most of the time, 5-always). The investigators will evaluate top-box (topmost, ie, "never") scores for this measure.
Safety Climate (The Children's Hospital Safety Climate Questionnaire) | 24 months (including usual care and intervention implementation data collection which will happen sequentially)per site (8 sites total)
  Self-reported by patients/families prior to discharge. The Children's Hospital Safety Climate Questionnaire includes 14 Likert-scale (agreement on a 5 point scale from "strongly agree" to "strongly disagree") questions related to parent perceptions of safety climate during hospitalization. It was adapted from the AHRQ Hospital Survey on Patient Safety Culture for staff and validated using confirmatory factor analysis. Domains include perceptions of safety, staff communication openness, parent communication openness, and handoffs and transitions. Items of interest relate to the communication openness domain. Top-box (top-most/best) scores will be analyzed.
Observations of Quality and Frequency of Communications | 24 months (including usual care and intervention implementation data collection which will happen sequentially) per site (8 sites total)
  Direct observations (by study staff) will measure the frequency of (1) overall communications between patients/families and providers, (2) language-concordant communications among patients and providers (times a provider communicates with a patient/family in a language the patient understands), and (3) interpreter-facilitated communications among patients with LEP. The type of communications and their quality will also be observed. The study team has used direct observations to measure frequency, type, and quality of communication reliably in multiple prior studies and will modify these prior measures to assess communication.

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Khan, MD, MPH, Principal Investigator — Boston Children's Hospital/Harvard Medical School
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital of Oakland, Oakland, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Children's Hospital at Montefiore, The Bronx, New York
  - The Research Institute of Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Northwest Texas Healthcare System, Amarillo, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Starmer AJ, Spector ND, Srivastava R, West DC, Rosenbluth G, Allen AD, Noble EL, Tse LL, Dalal AK, Keohane CA, Lipsitz SR, Rothschild JM, Wien MF, Yoon CS, Zigmont KR, Wilson KM, O'Toole JK, Solan LG, Aylor M, Bismilla Z, Coffey M, Mahant S, Blankenburg RL, Destino LA, Everhart JL, Patel SJ, Bale JF Jr, Spackman JB, Stevenson AT, Calaman S, Cole FS, Balmer DF, Hepps JH, Lopreiato JO, Yu CE, Sectish TC, Landrigan CP; I-PASS Study Group. Changes in medical errors after implementation of a handoff program. N Engl J Med. 2014 Nov 6;371(19):1803-12. doi: 10.1056/NEJMsa1405556. PMID 25372088
- [Background] Khan A, Coffey M, Litterer KP, Baird JD, Furtak SL, Garcia BM, Ashland MA, Calaman S, Kuzma NC, O'Toole JK, Patel A, Rosenbluth G, Destino LA, Everhart JL, Good BP, Hepps JH, Dalal AK, Lipsitz SR, Yoon CS, Zigmont KR, Srivastava R, Starmer AJ, Sectish TC, Spector ND, West DC, Landrigan CP; the Patient and Family Centered I-PASS Study Group; Allair BK, Alminde C, Alvarado-Little W, Atsatt M, Aylor ME, Bale JF Jr, Balmer D, Barton KT, Beck C, Bismilla Z, Blankenburg RL, Chandler D, Choudhary A, Christensen E, Coghlan-McDonald S, Cole FS, Corless E, Cray S, Da Silva R, Dahale D, Dreyer B, Growdon AS, Gubler L, Guiot A, Harris R, Haskell H, Kocolas I, Kruvand E, Lane MM, Langrish K, Ledford CJW, Lewis K, Lopreiato JO, Maloney CG, Mangan A, Markle P, Mendoza F, Micalizzi DA, Mittal V, Obermeyer M, O'Donnell KA, Ottolini M, Patel SJ, Pickler R, Rogers JE, Sanders LM, Sauder K, Shah SS, Sharma M, Simpkin A, Subramony A, Thompson ED Jr, Trueman L, Trujillo T, Turmelle MP, Warnick C, Welch C, White AJ, Wien MF, Winn AS, Wintch S, Wolf M, Yin HS, Yu CE. Families as Partners in Hospital Error and Adverse Event Surveillance. JAMA Pediatr. 2017 Apr 1;171(4):372-381. doi: 10.1001/jamapediatrics.2016.4812. PMID 28241211
- [Background] Khan A, Spector ND, Baird JD, Ashland M, Starmer AJ, Rosenbluth G, Garcia BM, Litterer KP, Rogers JE, Dalal AK, Lipsitz S, Yoon CS, Zigmont KR, Guiot A, O'Toole JK, Patel A, Bismilla Z, Coffey M, Langrish K, Blankenburg RL, Destino LA, Everhart JL, Good BP, Kocolas I, Srivastava R, Calaman S, Cray S, Kuzma N, Lewis K, Thompson ED, Hepps JH, Lopreiato JO, Yu CE, Haskell H, Kruvand E, Micalizzi DA, Alvarado-Little W, Dreyer BP, Yin HS, Subramony A, Patel SJ, Sectish TC, West DC, Landrigan CP. Patient safety after implementation of a coproduced family centered communication programme: multicenter before and after intervention study. BMJ. 2018 Dec 5;363:k4764. doi: 10.1136/bmj.k4764. PMID 30518517
- [Background] Khan A, Yin HS, Brach C, Graham DA, Ramotar MW, Williams DN, Spector N, Landrigan CP, Dreyer BP; Patient and Family Centered I-PASS Health Literacy Subcommittee. Association Between Parent Comfort With English and Adverse Events Among Hospitalized Children. JAMA Pediatr. 2020 Dec 1;174(12):e203215. doi: 10.1001/jamapediatrics.2020.3215. Epub 2020 Dec 7. PMID 33074313
- [Background] Parente VM, Khan A, Robles JM. Belonging on Rounds: Translating Research Into Inclusive Practices for Families With Limited English Proficiency to Promote Safety, Equity, and Quality. Hosp Pediatr. 2022 May 1;12(5):e171-e173. doi: 10.1542/hpeds.2022-006581. No abstract available. PMID 35411380
- [Background] Khan A, Quinones-Perez B, Castellanos A, Garcia S, MacInnes E. Promoting true meaningful access and equity for patients and clinicians through the use of certified interpreters in hospitals. J Hosp Med. 2022 Sep;17(9):772-773. doi: 10.1002/jhm.12943. Epub 2022 Aug 17. No abstract available. PMID 35977037
- [Background] Khan A, Parente V, Baird JD, Patel SJ, Cray S, Graham DA, Halley M, Johnson T, Knoebel E, Lewis KD, Liss I, Romano EM, Trivedi S, Spector ND, Landrigan CP; Patient and Family Centered I-PASS SCORE Scientific Oversight Committee; Bass EJ, Calaman S, Fegley AE, Knighton AJ, O'Toole JK, Sectish TC, Srivastava R, Starmer AJ, West DC. Association of Patient and Family Reports of Hospital Safety Climate With Language Proficiency in the US. JAMA Pediatr. 2022 Aug 1;176(8):776-786. doi: 10.1001/jamapediatrics.2022.1831. PMID 35696195